CLINICAL TRIAL: NCT01800188
Title: Glucose Metabolism During Hemodialysis
Status: Completed | Type: Observational
Sponsor: Bo Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, MD DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-2-2012-171
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: ESRD
Keywords: Dialysis; Incretin hormones
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis; Hemodiafiltration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum of blood specimens will be retained for analysis at the end of the study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dialysis: Patients with dialysis dependent ESRD and normal fasting glucose will undergo a meal test during a hemodialysis and hemodiafiltration session. A meal test without dialysis is optional.
  Interventions: Procedure: Hemodialysis; Procedure: Hemodiafiltration; Procedure: Meal test

INTERVENTIONS:
Procedure: Hemodialysis — A 4 hour hemodialysis with a standardized liquid meal after one hour
Procedure: Hemodiafiltration — A 4 hour hemodiafiltration with a standardized liquid meal after one hour
Procedure: Meal test — A 3 hour standardized liquid meal test without dialysis

SUMMARY:
Disturbed glucose metabolism is a common feature of patients with end-stage renal disease (ESRD). Several hormones responsible of a stable blood glucose including insulin, glucagon, and the gastrointestinal insulinotropic hormones Glucagon-like Peptide-1 (GLP-1) and Glucose-dependent Insulinotropic Peptide (GIP) are elevated in patients with ESRD. These hormones are all medium sized peptides which theoretically makes them removable during high efficient hemodialysis. A significant removal could have consequences for the treatment of patients with diabetes and ESRD.

The purpose of this study is to determine whether insulin, glucagon, GLP-1 and GIP are cleared during high efficient hemodialysis and hemodiafiltration. The investigators hypothesize that a significant amount of these hormones is removed during hemodialysis and to a larger extend during hemodiafiltration.

DETAILED DESCRIPTION:
BACKGROUND

Disturbed glucose metabolism is a common feature of patients with end-stage renal disease (ESRD). Furthermore, the prevalence of diabetes mellitus in the ESRD population is high resulting in a marked increased morbidity and mortality. Several hormones responsible of a stable blood glucose including insulin, glucagon, and the gastrointestinal insulinotropic hormones Glucagon-like Peptide-1 (GLP-1) and Glucose-dependent Insulinotropic Peptide (GIP) are elevated and dysregulated in patients with ESRD. Newly developed antidiabetic medications such as the dipeptidyl peptidase-4 inhibitors (DPP-4 inhibitors) increase the concentrations of these hormones making the effect of these treatments difficult to predict in patients with ESRD.

During the history of hemodialysis the treatment has been refined to increase the removal of the various substances that accumulate when the kidney function declines. The focus has primary been on the removal of smaller molecules such as creatinine and urea, but in recent decades the focus has moved to medium-sized molecules (molecular weight of 300 to 12,000 Da) which are suspected of causing various uremic complications such as amyloidosis and neuropathy. The dialysis technique has therefore been optimized such that relatively large molecules are removed, but the dialysis filter does not distinguish between wanted and unwanted substances. Thus, in contrast to the functioning kidney there is a risk of removing important molecules including hormones, which are essential for maintaining a normal glucose metabolism.

Insulin, glucagon and the incretin hormones, GLP-1 and GIP are all peptides with a molecular weight of 3300 to 5800 Da. This means that they theoretically have a size where they can be removed under hemodialysis with so-called high-flux filters and by hemodiafiltration, both of which are common standards of care for patients with ESRD. It has been shown that insulin is removed in significant quantities during a hemodialysis, but this is probably due to adsorption to the filter and not filtration. Whether glucagon and the incretin hormones are eliminated by high effective hemodialysis and hemodiafiltration is never investigated. Previous studies have primarily observed unchanged glucagon and GIP concentrations in the blood after conventional hemodialysis. One study showed a 30% decrease in GIP concentration after hemodialysis, but the detected change probably reflects altered metabolism due to the treatment as the dialysis technique at the time was too inefficient to remove peptides significantly. Assays for the analysis of incretin hormones have also become considerably more specific and now differentiate between the active hormones and their inactive intermediate metabolites.

In recent years there has been a growing development of drugs that increase the endogenous produced incretin hormones. Linagliptin, launched in 2011, is the only one that is approved for patients with ESRD since it is not cleared renally and therefore does not require a change in dosage. However, the elimination of incretin hormones in dialysis patients is sparingly studied both during and between dialysis treatments.

This study will determine the effect of high efficient dialysis treatment on a number of hormones regulating the blood glucose. Significant elimination of these hormones during dialysis can have therapeutic implications for the treatment of dialysis patients with incretin based therapies.

PURPOSE OF THE STUDY

The purpose of this study is to determine whether several blood glucose-regulating hormones and their metabolites are removed during hemodialysis and hemodiafiltration in patients with dialysis-dependent renal insufficiency. The hypothesis is that the dialysis treatment results in a significant removal, thereby reducing the plasma concentration of each hormone.

METHODS

10 patients with ESRD undergoing either chronic hemodialysis or chronic hemodiafiltration will be included. The study will be carried out on two separate days which are planned two days after their previous dialysis. On the two study days each participant will be treated with a 4 hour hemodialysis or hemodiafiltration. Besides the dialysis modality (hemodialysis and hemodiafiltration) the two study days will be alike.

The participant will be examined in the morning in a 10 hour fasting state (including smoking) without any alcohol consumption within the last 24 hours and strenuous physical activity within the last 2 hours. Weight, Height, blood pressure and pulse will be measured and the dialysis access is prepared. An initial blood sample will be analyzed immediately for sodium, bicarbonate and ionized calcium and the dialysate of the dialyzer will be adjusted to match the measured concentrations as close as possible. The ultrafiltration will be set according to the patients dry weight and no sodium or ultrafiltration profiles will be allowed. The blood flow will be held constant not exceeding the half of the flow of the arteriovenous fistula.

Each participant at each study day will receive the dialysis fasting for one hour after which a standardized liquid meal with 1.5 mg Paracetamol added will be administered.

During the dialysis blood samples will be measured repeatedly and analyzed for insulin, glucagon, GLP-1 and GIP. Blood samples will be drawn both before and after the dialysis filter to calculate the clearance and samples from the spend dialysate are collected to determine the amount of adsorption of the hormones to the dialysis filter.

Participants undergo an optional third examination day receiving the standardized meal test without dialysis. Blood samples are collected at the same time intervals as during the examination days with dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90 years
* Dialysis-dependent ESRD for more than 3 months
* Regular treatment with either hemodialysis or hemodiafiltration
* A well functioning arteriovenous fistula
* Fistula flow ≥ 400 ml/min

Exclusion Criteria:

* Diabetes mellitus
* Impaired fasting glucose (fasting plasma glucose ≥ 6.1 mmol/l)
* Current illness requiring admission to the hospital
* Significant acidosis before dialysis (standardized bicarbonate < 20 mmol/l)
* Anemia (B-Hemoglobin < 6,0 mmol/l)
* Known allergy to Paracetamol
* Medical treatment with compounds of known diabetogenic and / or insulin secretion inhibitory effect, including steroids and calcineurin inhibitors.
* Bowel resection or other major surgery of the gastrointestinal tract
* Current malignancy not including basal cell carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ESRD undergoing chronic hemodialysis/hemodiafiltration and with a normal fasting glucose
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Clearance of total GLP-1 | 2 hours into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.
Clearance of total GIP | 2 hours into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.
Clearance of glucagon | One hour into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.

SECONDARY OUTCOMES:
Change of insulin clearance at 2 hours into dialysis | Baseline and 2 hours into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.
Change of hormone concentrations | Baseline and 1 hour into dialysis
The percentage of cleared hormone present in the dialysate | One or two hours into the dialysis
Change of insulin clearance at 3 hours into dialysis | Baseline and 3 hours into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.
Change of insulin clearance at 4 hours into dialysis | Baseline and 4 hours into dialysis
  Clearance,K, is defined as
  K=Qb*(Ca-Cv)/Ca+Qf*Cv/Ca
  where Qb is the effective blood flow, Ca is the concentration before the filter, Cv is the concentration after the filter and Qf is the ultrafiltration flow.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, MD DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Nephrology department, Rigshospitalet, Copenhagen, Copenhagen, Denmark